CLINICAL TRIAL: NCT04479982
Title: Microbial Infections and Antimicrobial Resistance (AMR) Patterns Associated With Hospitalized Patients With 2019 Novel Coronavirus Disease (COVID 19)
Brief Title: Microbial Infection and AMR in Hospitalized Patients With Covid 19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ALShymaa faheem solyman ali, assistant lecturer, Assiut University
Other Study IDs: Microbial infection with covid
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To detect microbial infection and AMR associated with COVID 19 infection.

To correlate risk factors of COVID 19 patients with microbial infections and their effects on disease.

DETAILED DESCRIPTION:
The most common type of infection among ICU patients was bacterial or fungal pneumonia; bloodstream and urinary tract infections were also noted. Organisms cultured from patients included pandrug-resistant Acinetobacter baumannii, Klebsiella pneumoniae carbapenemase-producing K. pneumoniae, extended-spectrum β-lactamase (ESBL)- producing K. pneumoniae, ESBL-producing Pseudomonas aeruginosa, Enterobacter cloacae, Serratia marcescens, Aspergillus fumigatus, Aspergillus flavus, Candida albicans, and Candida glabrata .

ELIGIBILITY:
Inclusion Criteria:

* Patients with Covid infection

Exclusion Criteria:

* Patients without covid 19

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with covid 19
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-09-24 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbial infections and antimicrobial resistance (AMR) patterns associated with hospitalized patients with 2019 novel coronavirus disease (COVID 19) | baseline
  The correlation between microbial infection and COVID 19 infection and their effect on prognosis and disease outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut hopital, Asyut, Egypt